CLINICAL TRIAL: NCT02705183
Title: Post-operative RadioTherapy for Patients With Metastases of the Long Bones: a Randomised Controlled Trial
Brief Title: Post-operative RadioTherapy for Patients With Metastases of the Long Bones
Acronym: PORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, PD Sander Dijkstra, MD PhD, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL54480.058.15
Record Dates: First submitted 2016-02-25; First posted 2016-03-10 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Metastasis to Bone
Keywords: surgical treatment; post-operative radiotherapy; quality of life; complications; survival; long bones
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Surgery & Post-operative radiotherapy (Active Comparator): Surgery & Post-operative radiotherapy
  Interventions: Radiation: Radiotherapy
- B: Surgery only (No Intervention): Surgery only

INTERVENTIONS:
Radiation: Radiotherapy — Multifractionated post-operative radiotherapy, several weeks after surgery
  Arms: A: Surgery & Post-operative radiotherapy

SUMMARY:
Rationale: Bone metastases arise in 50% of all patients dying of cancer, increasing up to 70% in patients with breast and prostate cancer. The lesions can cause pain and fractures, leading to diminished quality of life and poorer survival. Current knowledge concerning adequate, personalized treatment of metastatic lesions of the long bones in patients with disseminated cancer is insufficient and inconclusive due to lack of large, prospective series with patient reported outcome measures. One of the debatable issues is the effectiveness of postoperative radiotherapy. It has become common practise due to professional opinion, but research evidence is lacking. It is thought that adjuvant radiotherapy improves the durability of an implant, prevents progression of the lesion, promotes bone healing, improves limb function, minimises pain and reduces the need for reoperations, however none of these are certain. Moreover, it is a burden on patient's quality of life (e.g. multiple extra hospital visits) causing toxicity and possible side effects (e.g. skin irritation). The true beneficial effect, weighing up the possible pros and certain cons, of adjuvant radiotherapy is thus unknown.

Objective: The PORT study aims to demonstrate the non-inferiority of 'surgery only' compared to surgery with adjuvant radiotherapy as treatment of impending and actual pathological fractures on the pain experienced by patients.

Study design: A multicentre, prospective, randomised non-inferiority trial nested within the OPTIMAL study.

Study population: All patients with metastases of the long bones undergoing surgery for a(n) (impending) pathologic fracture in the participating centres.

Study intervention: One study arm (A) will receive surgery with adjuvant radiotherapy; the other study arm (B) will receive surgery only.

Main study parameters/endpoints: Primary endpoint is patient reported pain according to a numeric rating scale (NRS). Clinical functioning, radiological status, complications and survival are secondary endpoints.

DETAILED DESCRIPTION:
The PORT study aims to demonstrate the non-inferiority of 'surgery only' compared to 'surgery with adjuvant radiotherapy' for the fixation of impending and actual pathological fractures of the long bones. We hypothesize that patients without post-operative radiotherapy will not have more pain than those receiving post-operative radiotherapy. The primary efficacy endpoint will be the pain level (as measured by an eleven point numeric rating scale (NRS)) 12 weeks after treatment. Pain has been chosen as primary endpoint because it can be interpreted as a "proxy" for mechanical loosening or other complications. It was undesirable to select revision surgery as endpoint, because the number of revision surgeries will be very low in this patient population. A revision will only be performed for serious complications with large effects on the quality of life. In other cases, conservative options will be chosen over revision surgery.

Secondary endpoints are complications, quality of life and overall survival.

A secondary objective is to conduct cost-effectiveness and costs-utility analyses.

This study is a multicentre, prospective, randomised non-inferiority trial nested within the OPTIMAL study. The OPTIMAL study is the backbone of the (OPTIMAL-) PORT study, encompassing the prospective cohort and providing the infrastructure for collection patient reported outcome measures. If patients do not have an indication for surgery, they can only be included in the OPTIMAL study. If patients have an indication for surgery, they are recruited for the OPTIMAL-PORT study. However, if patients do not give consent for randomisation for radiotherapy, they can give partial consent and participate in the prospective cohort and complete questionnaires. This data will contribute to the OPTIMAL study. Details concerning the OPTIMAL study are described in the respective protocol.

The PORT trial is a non-inferiority trial between ' surgery with post-operative radiotherapy' (Arm A) with 'surgery only (no post-operative radiotherapy)' (Arm B). A non-inferiority design is appropriate for this study because we expect that the clinical outcomes with surgery only are not worse than with post-operative radiotherapy. 'Surgery only' however has evident advantages, as it will lessen the burden on patients of visiting the hospital, prevent toxicity and cost less. Furthermore, as mentioned in the introduction, the focus of treatment is on maintaining and improving quality of life. The goal is to do what is right, safe, and efficient and not to provide more care than is needed. Rethinking whether we need post-operative radiotherapy is part of achieving that goal.

All patients with (impending) fractures of the long bones due to bone metastases and an operation indication will be asked to participate in the OPTIMAL cohort and provide patient reported outcomes. In addition, they will be informed about the PORT trial. Post-operatively, shortly before discharge from the hospital, they will be asked for informed consent for the PORT trial by the treating physician or a researcher. This assures a waiting period of 3-7 days between information and consent. Patients are informed that they are free to decide whether they wish to participate in the trial and will receive written information in addition to oral information. If patients do not wish to participate in the trial, they will receive standard care (which is post-operative radiotherapy in most cases). The first post-operative questionnaire will be sent 4 weeks after surgery.

Statistical analysis: To describe patient characteristics and outcomes, descriptive statistics (mean, median, standard deviation, and proportions) will be used. For univariate testing, p-values will be one tailed and considered significant if less than 0.05.

The primary endpoint of this study is pain response after surgery with or without post-operative radiotherapy. This will be expressed in absolute numbers (difference in NRS). A linear regression model to adjust for patients' characteristics will be used to compare the difference in mean pain level between the two arms with the centre from which the patient originates as a random effect.

For the analysis of non-inferiority primarily an intention to treat (ITT) will be performed. However, an ITT analysis is more likely to narrow the difference between treatments in a non-inferiority trial and yield a non-inferior result, thus a per protocol (PP) analysis is needed to cross-validate the ITT analysis.

Differences in the occurrence of complications will be compared by Fisher's exact test or chi-square test.

The QoL will be analysed using the EORTC QLQ-C15-PAL and EORTC QLQ-BM22. A comparison will be made between the baseline QoL and at predefined intervals after treatment (at 4 and 8 weeks, 3, 6 and 12 months following radiotherapy). A change of 10% of the scale width will be considered a clinically relevant change of QoL (Osoba 2005). The data will be presented as stable, worsened (≥ 10% decrease in QoL) or improved (≥ 10%increase in QOL). These time points will be compared using a Chi square test with a conservative p-value of 0.01 to correct for multiple testing. We will also evaluate the pattern of QoL as a continuous outcome over time during follow up with the mixed models approach.

Overall survival and progression free survival will be estimated by applying Kaplan-Meier's methodology analysis. Time to event will be measured from time of treatment to death or to progression of the disease. Comparisons in outcomes between treatment groups will be performed by Log Rank test.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Bone metastasis deriving from the following bones:

  * humerus, ulna, radius
  * femur, tibia, fibula
* Radiographic or histologic proof of metastatic bone disease
* Histologic diagnosis of the primary tumour or - if the diagnosis is unknown - at least adequate diagnostic investigations into the origin of the metastasis (e.g. dissemination imaging, histology, biopsy)
* Receive surgical treatment with palliative intent for a pathologic fracture or impending pathologic fracture

Exclusion Criteria:

* Primary bone tumours (benign and/or malignant)
* No informed consent signed
* Communication with patient is hampered (e.g. language barrier, severe cognitive impairment, dementia)
* Lesions in the small bones of the extremities
* (Surgical) treatment with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with a difference of 2 points or more on a 11-point numeric rating scale for pain | 3 months
  Pain will measured before treatment and after treatment on an 11-point numeric rating scale for pain. If the score differs more than 2 points between those measuring moments the change in pain is reported as significant. The number of patients in each group with a significant change in pain score will be measured.

SECONDARY OUTCOMES:
Complications | 3 months, 6 months, 1 year
  Complications such as loosening of implant

CONTACTS AND LOCATIONS:
Overall Officials: Sander Dijkstra, MD PhD, Principal Investigator — Leiden University Medical Center; Yvette van der Linden, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of OPTIMAL Study, including PORT study — http://www.optimal-study.nl